CLINICAL TRIAL: NCT04363801
Title: A Phase 2, Multicenter, Open-Label Study of DKN-01 in Combination With Tislelizumab ± Chemotherapy as First-Line or Second-Line Therapy in Adult Patients With Inoperable, Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma (DisTinGuish)
Brief Title: A Study of DKN-01 in Combination With Tislelizumab ± Chemotherapy in Patients With Gastric or Gastroesophageal Cancer
Acronym: DisTinGuish
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: experimental treatment will not be more efficacious than its comparator in the primary endpoint of PFS
Sponsor: Leap Therapeutics, Inc. (Industry)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEK-DKK1-P205
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma; GastroEsophageal Cancer
Keywords: Gastric cancer; Gastroesophageal junction; cancer; adenocarcinoma; DKK1; Tislelizumab; DKN-01
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms; Adenocarcinoma | interventions — tislelizumab; Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A First Line Treatment (Experimental): Part A patients will receive IV DKN-01 (300 mg) on Days 1 and 15, IV tislelizumab (200 mg) on Day 1, IV oxaliplatin (130 mg/m2) on Day 1, and oral capecitabine (1000 mg/m2 twice daily [BID]) on Days 1-15 of each 21-day cycle. Part A is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  Interventions: Drug: DKN-01 300mg; Drug: DKN-01 400mg; Drug: Tislelizumab 200mg; Drug: Tislelizumab 400mg
- Part B1 Second Line Treatment (Experimental): Part B patients will receive IV DKN-01 (300 mg) on Days 1 and 15 and IV tislelizumab (200 mg) on Day 1 of each 21-day cycle.
  Patients enrolled in Part B are required to have DKK1-high (H-score ≥ 35) G/GEJ adenocarcinoma (pre-screen biopsy) and must have had only 1 prior systemic therapy for locally advanced/metastatic disease (platinum + fluoropyrimidine-based therapy; ±Human Epidermal growth factor Receptor 2 [HER2] therapy if applicable). Patients may have received prior neoadjuvant or adjuvant therapy.
  Interventions: Drug: DKN-01 300mg; Drug: DKN-01 400mg
- Part B2 Second Line Treatment (Experimental): Part B patients will receive IV DKN-01 (600 mg) on Days 1 and 15 and IV tislelizumab (200 mg) on Day 1 of each 21-day cycle.
  Patients enrolled in Part B are required to have DKK1-high (H-score ≥ 35) G/GEJ adenocarcinoma (pre-screen biopsy) and must have had only 1 prior systemic therapy for locally advanced/metastatic disease (platinum + fluoropyrimidine-based therapy; ±HER2 therapy if applicable). Patients may have received prior neoadjuvant or adjuvant therapy.
  Interventions: Drug: DKN-01 600mg; Drug: DKN-01 400mg
- Part C Control First Line Treatment (Active Comparator): Part C control patients will receive only tislelizumab in combination with chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  Interventions: Drug: Tislelizumab 200mg; Drug: Tislelizumab 400mg; Drug: Oxaliplatin; Drug: Capecitabine 1000mg/ m2 twice daily (BID); Drug: Leucovorin Calcium; Drug: Fluorouracil
- Part C Experimental First Line Treatment (Experimental): Part C experimental patients will receive DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  Interventions: Drug: DKN-01 600mg; Drug: DKN-01 400mg; Drug: Tislelizumab 200mg; Drug: Tislelizumab 400mg; Drug: Oxaliplatin; Drug: Capecitabine 1000mg/ m2 twice daily (BID); Drug: Leucovorin Calcium; Drug: Fluorouracil

INTERVENTIONS:
Drug: DKN-01 300mg — Administered by IV infusion
  Other Names: Experimental
  Arms: Part A First Line Treatment; Part B1 Second Line Treatment
Drug: DKN-01 600mg — Administered by IV infusion
  Other Names: Experimental
  Arms: Part B2 Second Line Treatment; Part C Experimental First Line Treatment
Drug: DKN-01 400mg — Administered by IV infusion
  Other Names: Experimental
  Arms: Part A First Line Treatment; Part B1 Second Line Treatment; Part B2 Second Line Treatment; Part C Experimental First Line Treatment
Drug: Tislelizumab 200mg — Administered by IV infusion
  Other Names: humanized IgG4 anti-PD-1 monoclonal antibody; Tevimbra
  Arms: Part A First Line Treatment; Part C Control First Line Treatment; Part C Experimental First Line Treatment
Drug: Tislelizumab 400mg — Administered by IV infusion
  Other Names: humanized IgG4 anti-PD-1 monoclonal antibody; Tevimbra
  Arms: Part A First Line Treatment; Part C Control First Line Treatment; Part C Experimental First Line Treatment
Drug: Oxaliplatin — Administered by IV infusion
  Other Names: Eloxatin
  Arms: Part C Control First Line Treatment; Part C Experimental First Line Treatment
Drug: Capecitabine 1000mg/ m2 twice daily (BID) — Administered orally
  Other Names: Xeloda
  Arms: Part C Control First Line Treatment; Part C Experimental First Line Treatment
Drug: Leucovorin Calcium — Administered by IV infusion
  Other Names: Folinic acid
  Arms: Part C Control First Line Treatment; Part C Experimental First Line Treatment
Drug: Fluorouracil — Administered by IV infusion
  Other Names: 5-FU
  Arms: Part C Control First Line Treatment; Part C Experimental First Line Treatment

SUMMARY:
A Phase 2, Multicenter, Open-Label Study of DKN-01 in Combination with Tislelizumab ± Chemotherapy as First-Line or Second-Line Therapy in Adult Patients with Inoperable, Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma

DETAILED DESCRIPTION:
This is a Phase 2 open-label, multicenter study to be conducted concurrently in 3 Parts (Parts A, B, and C). Approximately 232 patients aged 18 years or older with inoperable, histologically confirmed locally advanced or metastatic Gastric or Gastroesophageal Junction (G/GEJ) adenocarcinoma with measurable disease (RECIST v1.1) requiring therapy will be enrolled in the study. Part A and B are designed to evaluate safety, tolerability, and efficacy of the combination therapy of intravenous (IV) DKN-01 and tislelizumab ± CAPOX in G/GEJ adenocarcinoma patients. Treatment continues in repeating 21-day cycles until patient meets criteria for discontinuation or is no longer deriving clinical benefit. Two doses of DKN-01 will be evaluated in Part B (Part B1 and Part B2). Part C is the open-label, randomized, controlled, 2-arm portion of the study to evaluate the efficacy and safety of tislelizumab + chemotherapy regimen (CAPOX or mFOLFOX6) ± DKN-01 in adult patients with inoperable, histologically confirmed locally advanced or metastatic G/GEJ adenocarcinoma with measurable disease (RECIST v1.1) requiring therapy. Approximately 160 patients will be randomized in a 1:1 ratio to receive either DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6) (n=80) or tislelizumab in combination with chemotherapy regimen (CAPOX or mFOLFOX6) (n=80).

ELIGIBILITY:
Inclusion:

Part A & C:

1. No previous therapy for cancer. Patients may have received prior neoadjuvant or adjuvant therapy as long it was completed without disease recurrence for at least 6 months since last treatment.

   Part B Only:
2. Disease progression during first-line therapy or within 4 months after the last dose of first-line therapy.
3. Documentation of elevated Dickkopf-1 (DKK1) messenger ribonucleic acid (mRNA) expression from a fresh tumor biopsy or a biopsy obtained within the 6 months of screening.

   Part C Only:
4. Documentation of programmed cell death protein ligand-1 (PD-L1) combined positive score (CPS) by immunohistochemistry (IHC) and DKK1 mRNA expression in tumor cells by ISH from a fresh tumor biopsy (preferred) or archived tumor biopsy specimen conducted in a Sponsor designated central laboratory.

   General:
5. Able to provide written informed consent prior to any study-specific procedures.
6. Age ≥18 years on the day of signing the informed consent (exception: ≥19 years in the Republic of Korea).
7. Confirmed diagnosis of gastric adenocarcinoma or gastroesophageal junction (GEJ) adenocarcinoma.
8. One or more tumors measurable on radiographic imaging as defined by Response Evaluation Criteria in Solid Tumor (RECIST) 1.1.
9. Tumor tissue for mandatory pre-treatment evaluation (fresh biopsy [preferred] or archived specimen).
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 within 7 days of first dose of study drug
11. Acceptable liver, renal, hematologic, and coagulation function
12. Females of childbearing potential and male partners of female patients must agree to use adequate contraception during the study and for 6 months after their last dose of study drug.
13. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for at least 6 months after the last dose of study drugs.

Exclusion:

Part A & C Only:

1. Diagnosis of HER2-positive G/GEJ adenocarcinoma.
2. Unable to swallow capsules or disease significantly affected gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction (for those receiving CAPOX in Part C).
3. Prior therapy with an anti-programmed cell death protein 1 (PD-1) or anti-PD-L1 antibody.

   Part B Only:
4. Major surgery or chemotherapy within 21 days of first dose of study drug.

   General:
5. Squamous cell or undifferentiated or other histological type of gastric cancer.
6. Prior therapy with an anti-PD-L2 or any other antibody or drug specifically targeting T-cell co-stimulation or co-inhibitory checkpoint pathways in any treatment setting (including adjuvant/neoadjuvant) or prior therapy with an anti-DKK1 agent.
7. Patients with active autoimmune diseases or history of autoimmune diseases that may relapse.
8. Any condition that required treatment with steroids or any other immune suppressive drugs within 14 days prior to first dose of study drug.
9. Active leptomeningeal disease or uncontrolled brain metastases.
10. Any active cancer ≤ 2 years before first dose of study drug with the exception of cancer for this study.
11. Uncontrolled diabetes or >Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management or ≥Grade 3 hypoalbuminemia within 14 days before first dose of study drug.
12. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage within 7 days prior to first dose of study drug.
13. Clinically significant anorexia within 7 days prior to first dose of study drug.
14. History of interstitial lung disease, non-infectious pneumonitis, pulmonary fibrosis, acute lung disease, or uncontrolled systemic diseases.
15. Active, uncontrolled bacterial, viral, or fungal infections, within 14 days of study entry requiring systemic therapy.
16. Prior allogeneic stem cell transplantation or organ transplantation.
17. History of severe hypersensitivity reactions to other monoclonal antibodies or any components of study treatment.
18. Known dihydropyrimidine dehydrogenase deficiency.
19. New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, or unstable arrhythmia.
20. Fridericia-corrected QT interval (QTcF) > 470 msec (female) or history of congenital long QT syndrome.
21. Known to be human immunodeficiency virus (HIV) positive.
22. Serious nonmalignant disease
23. History of osteonecrosis of the hip or have evidence of structural bone abnormalities in the proximal femur on magnetic resonance imaging (MRI) scan that are symptomatic and clinically significant.
24. Known osteoblastic bony metastasis.
25. History of gastrointestinal perforation and/or fistulae within 6 months prior to first dose of study drug.
26. Major surgery 28 days prior to study entry.
27. Serious psychiatric or medical conditions that could interfere with treatment.
28. Toxicities (as a result of prior anticancer therapy) that have not recovered to baseline or stabilized, except for Adverse Events (AEs) not considered a likely safety risk (e.g., alopecia, neuropathy, and specific laboratory abnormalities).
29. Administration of a live vaccine within 28 days before first dose of study drug.
30. Active substance abuse.
31. Pregnant or nursing.
32. Concurrent participation in another therapeutic clinical study.
33. Prior radiation therapy within 14 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Sirard, MD, Study Director — Chief Medical Officer
Locations (48):
- United States (23):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - City of Hope, Duarte, California
  - The Angeles Clinic Research Institute - A Cedars-Sinai Affiliate, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - UCLA, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California
  - University of California San Francisco, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Germany (7):
  - Charité Universitätsmedizin Berlin, Berlin
  - Institut Fur Klinisch Onkologische Forschung Am Krankenhaus Nordwest, Frankfurt
  - Hämatologisch-Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Slk-Kliniken, Heilbronn
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Caritas Klinikum Saarbrücken St. Theresia, Saarbrücken
- South Korea (18):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Korea University Ansan Hospital, Ansan-si
  - Hallym University Sacred Heart Hospital, Anyang
  - Dong-A University Hospital, Busan
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Boramae Hospital SNU, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea St. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon

REFERENCES:
- [Derived] Klempner SJ, Sonbol MB, Wainberg ZA, Uronis HE, Chiu VK, Scott AJ, Iqbal S, Tejani MA, Chung V, Stilian MC, Thoma M, Zhang Y, Kagey MH, Baum J, Sirard CA, Altura RA, Ajani JA. DKN-01 in Combination With Tislelizumab and Chemotherapy as First-Line Therapy in Advanced Gastric or Gastroesophageal Junction Adenocarcinoma: DisTinGuish. J Clin Oncol. 2025 Jan 20;43(3):339-349. doi: 10.1200/JCO.24.00410. Epub 2024 Oct 21. PMID 39432867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2 open-label, multicenter study conducted concurrently in 3 parts: Non-randomized Parts A and B, and a randomized Part C.
Groups:
- Part B1 Second Line Treatment: Part B patients will receive IV DKN-01 (300 mg) on Days 1 and 15 and IV tislelizumab (200 mg) on Day 1 of each 21-day cycle.
  Patients enrolled in Part B are required to have Dickkopf-1 (DKK1)-high (H-score ≥ 35) gastric or gastroesophageal junction (G/GEJ) adenocarcinoma (pre-screen biopsy) and must have had only 1 prior systemic therapy for locally advanced/metastatic disease (platinum + fluoropyrimidine-based therapy; ±human epidermal growth factor receptor 2 (HER2) therapy if applicable). Patients may have received prior neoadjuvant or adjuvant therapy.
  DKN-01 300mg: Administered by IV infusion
  DKN-01 400mg: Administered by IV infusion
- Part B2 Second Line Treatment: Part B patients will receive IV DKN-01 (600 mg) on Days 1 and 15 and IV tislelizumab (200 mg) on Day 1 of each 21-day cycle.
  Patients enrolled in Part B are required to have DKK1-high (H-score ≥ 35) G/GEJ adenocarcinoma (pre-screen biopsy) and must have had only 1 prior systemic therapy for locally advanced/metastatic disease (platinum + fluoropyrimidine-based therapy; ±HER2 therapy if applicable). Patients may have received prior neoadjuvant or adjuvant therapy.
  DKN-01 600mg: Administered by IV infusion
  DKN-01 400mg: Administered by IV infusion
- Part C Control First Line Treatment: Part C control patients will receive only tislelizumab in combination with chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  Tislelizumab 200mg: Administered by IV infusion
  Tislelizumab 400mg: Administered by IV infusion
  Oxaliplatin: Administered by IV infusion
  Capecitabine 1000mg/ m2 BID: Administered orally
  Leucovorin Calcium: Administered by IV infusion
  Fluorouracil: Administered by IV infusion
- Part C Experimental First Line Treatment: Part C experimental patients will receive DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  DKN-01 600mg: Administered by IV infusion
  DKN-01 400mg: Administered by IV infusion
  Tislelizumab 200mg: Administered by IV infusion
  Tislelizumab 400mg: Administered by IV infusion
  Oxaliplatin: Administered by IV infusion
  Capecitabine 1000mg/ m2 BID: Administered orally
  Leucovorin Calcium: Administered by IV infusion
  Fluorouracil: Administered by IV infusion
Period: Overall Study
Arm/Group | Part A First Line Treatment | Part B1 Second Line Treatment | Part B2 Second Line Treatment | Part C Control First Line Treatment | Part C Experimental First Line Treatment
Started | 25 | 24 | 28 | 85 | 85
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 25 | 24 | 28 | 85 | 85
Not completed — Death | 18 | 14 | 16 | 48 | 38
Not completed — Withdrawal by Subject | 1 | 6 | 1 | 4 | 14
Not completed — Sponsor Decision | 6 | 4 | 10 | 33 | 32
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Parts A & B planned for 72 subjects enrolled: 25 subjects enrolled in Part A, 53 subjects enrolled in Part B. The Safety population consisted of 25 subjects in Part A, 52 subjects in Part B; the modified Intent-to-Treat population consisted of 22 subjects in Part A, 52 patients in Part B. Part C planned for 160 subjects enrolled: 170 subjects were randomized, with 84 treated subjects in the experimental group, 85 treated subjects in the control group.
Groups:
- Part B1 Second Line Treatment: Part B patients will receive IV DKN-01 (300 mg) on Days 1 and 15 and IV tislelizumab (200 mg) on Day 1 of each 21-day cycle.
  Patients enrolled in Part B are required to have DKK1-high (H-score ≥ 35) G/GEJ adenocarcinoma (pre-screen biopsy) and must have had only 1 prior systemic therapy for locally advanced/metastatic disease (platinum + fluoropyrimidine-based therapy; ±HER2 therapy if applicable). Patients may have received prior neoadjuvant or adjuvant therapy.
  DKN-01 300mg: Administered by IV infusion
  DKN-01 400mg: Administered by IV infusion
- Total: Total of all reporting groups
Arm/Group | Part A First Line Treatment | Part B1 Second Line Treatment | Part B2 Second Line Treatment | Part C Control First Line Treatment | Part C Experimental First Line Treatment | Total
Number analyzed (Participants) | 25 | 24 | 28 | 85 | 85 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 16 | 50 | 57 | 154
  >=65 years | 9 | 9 | 12 | 35 | 28 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.65) | 59.0 (7.94) | 60.0 (13.70) | 59.8 (12.76) | 59.0 (11.39) | 59.4 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 7 | 21 | 26 | 64
  Male | 19 | 20 | 21 | 64 | 59 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 5 | 1 | 12
  Not Hispanic or Latino | 22 | 22 | 26 | 80 | 82 | 232
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 14 | 18 | 54 | 51 | 138
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 2 | 3
  White | 20 | 9 | 9 | 28 | 30 | 96
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 1 | 3 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants] — 25 patients from the USA were enrolled in Part A, and 53 patients from the USA and The Republic of South Korea were enrolled in Part B. The Safety population consisted of 25 patients in Part A and 52 patients in Part B, and the modified Intent-to-Treat (mITT) population consisted of 22 patients in Part A and 52 patients in Part B.
  In Part C, 170 patients were randomized from the USA, The Republic of South Korea, and Germany. The Safety population consisted of 169 patients and the Intent-to-Treat (ITT) population consisted of 170 patients. Population: Descriptive statistics were used to summarize demographics and Baseline characteristics for the Safety and mITT populations. In addition, select Baseline characteristics were analyzed with respect to geographic region, i.e., USA versus The Republic of South Korea.
  Participants
    South Korea | 0 | 14 | 16 | 51 | 49 | 130
    United States | 25 | 10 | 12 | 30 | 30 | 107
    Germany | 0 | 0 | 0 | 4 | 6 | 10
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: Some subject data in Part C not available for analysis of BSA
  m^2
    number analyzed (Participants) | 25 | 24 | 28 | 83 | 84 | 244
    (all) | 2.0 (0.23) | 1.8 (0.25) | 1.8 (0.26) | 1.8 (0.25) | 1.8 (0.28) | 1.8 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Part A and B: Safety and Tolerability of DKN-01 in G/GEJ Patients
Description: Number of subjects with adverse drug reactions and toxicities as assessed by CTCAE v5.0 CAPOX (capecitabine + oxaliplatin) in patients with inoperable, locally advanced or metastatic G/GEJ adenocarcinoma.
Time Frame: approximately 28 months
Population: In Parts A and B, 25 patients were enrolled in Part A and 53 patients were enrolled in Part B. The Safety population consisted of 25 patients in Part A and 52 patients in Part B, and the modified Intent-to-Treat (mITT) population consisted of 22 patients in Part A and 52 patients in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A First Line Treatment | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 25 | 24 | 28
Participants | 25 | 24 | 25

2. Primary Outcome: Part C: Progression Free Survival (PFS) in G/GEJ DKK1 High and Overall Patients Treated With DKN-01 in Combination With Tislelizumab and Chemotherapy vs Tislelizumab and Chemotherapy as a First-line Therapy
Description: PFS was measured from the date of randomization to the date of documented disease progression, based on investigator assessed radiologic review using RECIST v1.1, or death due to any cause, whichever occurred first. If the patient had not died, but there was no radiographic post-baseline tumor assessment, PFS was censored at the date of randomization. If there were radiographic post-baseline tumor assessments that verified lack of disease progression, PFS was censored at the most recent tumor assessment before the data cut-off or study withdrawal, whichever occurred first.
Time Frame: approximately 30 months
Population: Experimental group: Sirexatamab + tislelizumab + CAPOX/FOLFOX; Control group: Tislelizumab + CAPOX/FOLFOX
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part C Control First Line Treatment | Part C Experimental First Line Treatment
Number analyzed (Participants) | 85 | 85
Months | 10.41 [7.75 to 13.86] | 7.66 [6.87 to 9.49]
Statistical Analysis 1: Comparison: Part C Control First Line Treatment vs Part C Experimental First Line Treatment; Test type: Superiority; p = 0.9676, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.98 to 2.05]

3. Secondary Outcome: Part A: Objective Response Rate (ORR) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab + CAPOX as a First-line Therapy
Description: Objective Response Rate (ORR) is defined as the proportion of patients achieving best overall response of Complete Response (CR) or Partial Response (PR) through radiological assessment of tumor response, based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Investigators were urged to have the same radiographic imaging modality used throughout the study for each subject (at baseline and at subsequent assessments) in order to provide uniformity of radiographic assessments.
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 22
percentage of patients | 72.7 [49.8 to 89.3]

4. Secondary Outcome: Part B: Objective Response Rate (ORR) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: Objective Response Rate (ORR) is defined as the proportion of patients achieving best overall response of Complete Response (CR) or Partial Response (PR) as assessed with Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 22 | 24
percentage of patients | 18.2 [5.19 to 40.3] | 25.0 [9.77 to 46.7]

5. Secondary Outcome: Part A: Duration of Response (DoR) in G/GEJ Patients Treated With DKN-01 With Tislelizumab + CAPOX as a First-line Therapy
Description: DoR is defined only for responders (patients with BOR of CR or PR) as the time from initial response until radiographically documented progressive disease or death due to any cause, whichever is earlier.
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01. Patients who do not experience PD or death at the time of the analysis were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 16
months | 10.0 [5.1 to 19.2]

6. Secondary Outcome: Part A: Duration of Complete Response (DoCR) in G/GEJ Patients Treated With DKN-01 With Tislelizumab + CAPOX as a First-line Therapy
Description: DoCR is defined as the time from initial complete response (CR) until radiographically documented progressive disease or death due to any cause, whichever is first.
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 1
months | 12.7 [NA to NA] — 95% Confidence Interval not calculable for a single participant

7. Secondary Outcome: Part A: Progression Free Survival (PFS) in G/GEJ Patients Treated With DKN-01 With Tislelizumab + CAPOX as a First-line Therapy
Description: For RECIST, PFS is defined as the time from first study drug dose (i.e., C1D1) to first radiographically documented progressive disease or death due to any cause.
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 22
Months | 11.8 [7.9 to NA] — The upper confidence limit (UCL) for the 50th percentile is defined as the first time at which the UCL for S(t) (based on a ln(-lnS(t)) transformation) is less than or equal too 1-50/100=0.5. There is never an observed failure time for which the upper bound of the confidence interval (CI) for the Kaplan Meier (KM) estimate (calculated using the Greenwood's method, different from ln(-lnS(t)) transformation) is less than 0.5, due to lack of events & sample size.

8. Secondary Outcome: Part A: Overall Survival (OS) in G/GEJ Patients Treated With DKN-01 With Tislelizumab + CAPOX as a First-line Therapy
Description: Overall survival (OS) is defined as the time from first study drug dose (i.e., C1D1) to first radiographically documented progressive disease or death due to any cause.
Time Frame: approximately 28 months
Population: The mITT population is defined as all patients who received more than one dose of DKN-01.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 22
months | 19.7 [15.3 to NA] — The upper confidence limit for the 50th percentile is defined as the first time at which the upper confidence limit for S(t) (based on a ln(-lnS(t)) transformation) is less than or equal to 1-50/100 =0.5. There is never an observed failure time for which the upper bound of the confidence interval for the KM estimate (calculated using the Greenwood's method, which is different from the ln(-lnS(t)) transformation above) is less than 0.5, due to lack of events and sample size.

9. Secondary Outcome: Part A: Duration of Clinical Benefit (DoCB) in G/GEJ Patients Treated With DKN-01 With Tislelizumab + CAPOX as a First-line Therapy
Description: DoCB is defined as the time from the initiation of DKN-01 to the time of progressive disease or death due to any cause, whichever occurs first, for patients who had a BOR of CR, PR, or SD of ≥6 weeks.
Time Frame: approximately 28 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 20
months | 11.9 [8.2 to NA] — The upper confidence limit for the 50th percentile is defined as the first time at which the upper confidence limit for S(t) (based on a ln(-lnS(t)) transformation) is less than or equal to 1-50/100 =0.5. There is never an observed failure time for which the upper bound of the confidence interval for the KM estimate (calculated using the Greenwood's method, which is different from the ln(-lnS(t)) transformation above) is less than 0.5, due to lack of events and sample size.

10. Secondary Outcome: Part A: Durable Clinical Benefit (DCB) in G/GEJ Patients Treated With DKN-01 With Tislelizumab + CAPOX as a First-line Therapy
Description: Durable clinical benefit (DCB) is defined as the proportion of patients presenting a Duration of clinical benefit (DoCB) for ≥180 days from initiation of DKN-01. Patients who have a best overall response of PD or those with clinical benefit lasting <180 days are not included.
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 22
percentage of patients | 72.7 [49.8 to 89.3]

11. Secondary Outcome: Part A: Disease Control Rate (DCR) in G/GEJ Patients Treated With DKN-01 With Tislelizumab + CAPOX as a First-line Therapy
Description: DCR is defined as the proportion of patients presenting with a best overall response (BOR) of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) for a duration of at least 6 weeks from initiation of DKN-01, as assessed by the Investigator using RECIST v1.1.
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part A First Line Treatment
Number analyzed (Participants) | 22
percentage of patients | 95.5 [77.2 to 99.9]

12. Secondary Outcome: Part B: Duration of Response (DoR) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: as for outcome 5
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01. Patients who do not experience progressive disease (PD) or death at the time of the analysis were censored. The median DoR was not reached in the 300 mg dose group.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part B1 Second Line Treatment: Patients will receive IV DKN-01 (300 mg) on Days 1 and 15 and IV tislelizumab (200 mg) on Day 1 of each 21-day cycle.
  Patients enrolled in Part B are required to have DKK1-high (H-score ≥ 35) G/GEJ adenocarcinoma (pre-screen biopsy) and must have had only 1 prior systemic therapy for locally advanced/metastatic disease (platinum + fluoropyrimidine-based therapy; ±HER2 therapy if applicable). Patients may have received prior neoadjuvant or adjuvant therapy.
  DKN-01 300mg: Administered by IV infusion
  DKN-01 400mg: Administered by IV infusion
- Part B2 Second Line Treatment: Patients will receive IV DKN-01 (600 mg) on Days 1 and 15 and IV tislelizumab (200 mg) on Day 1 of each 21-day cycle.
  Patients enrolled in Part B are required to have DKK1-high (H-score ≥ 35) G/GEJ adenocarcinoma (pre-screen biopsy) and must have had only 1 prior systemic therapy for locally advanced/metastatic disease (platinum + fluoropyrimidine-based therapy; ±HER2 therapy if applicable). Patients may have received prior neoadjuvant or adjuvant therapy.
  DKN-01 600mg: Administered by IV infusion
  DKN-01 400mg: Administered by IV infusion
Arm/Group | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 4 | 6
months | NA [1.5 to NA] — insufficient number of participants with events | 5.6 [2.3 to NA] — insufficient number of participants with events

13. Secondary Outcome: Part B: Duration of Complete Response (DoCR) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: Duration of complete response (DoCR) is defined as the time from initial CR until radiographically documented progressive disease or death due to any cause, whichever is first. No patients had a complete response (CR); therefore, the DoCR was not applicable.
Time Frame: approximately 28 months
Reporting Status: Not Posted

14. Secondary Outcome: Part B: Progression Free Survival (PFS) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: as for outcome 7
Time Frame: approximately 28 months
Population: The mITT population is defined as all patients who received more than one dose of DKN-01.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 22 | 24
months | 1.4 [1.3 to 2.3] | 1.4 [1.2 to 6.8]

15. Secondary Outcome: Part B: Overall Survival (OS) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: as for outcome 8
Time Frame: approximately 28 months
Population: The mITT population is defined as all patients who received more than one dose of DKN-01.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 22 | 24
months | 8.2 [2.6 to 18.0] | 7.7 [3.8 to NA] — insufficient number of participants with events

16. Secondary Outcome: Part B: Duration of Clinical Benefit (DoCB) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: Duration of clinical benefit (DoCB) is defined as the time from the initiation of DKN-01 to the time of progressive disease or death due to any cause, whichever occurs first, for patients who had a BOR of CR, PR, or SD of ≥6 weeks.
Time Frame: approximately 28 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 4 | 8
months | NA [11.8 to NA] — insufficient number of participants with events | NA [6.8 to NA] — insufficient number of participants with events

17. Secondary Outcome: Part B: Durable Clinical Benefit (DCB) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: DCB rate is defined as the proportion of patients presenting a DoCB (Duration of clinical benefit) for ≥ 180 days from initiation of DKN-01, Patients who have a best overall response of PD or those with clinical benefit lasting <180 days will not be included.
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 22 | 24
percentage of patients | 18.2 [5.19 to 40.3] | 33.3 [15.6 to 55.3]

18. Secondary Outcome: Part B: Disease Control Rate (DCR) in G/GEJ Patients Treated With DKN-01 in Combination With Tislelizumab as a Second-line Therapy
Description: as for outcome 11
Time Frame: approximately 28 months
Population: The modified Intent-to-Treat (mITT) population is defined as all patients who received more than one dose of DKN-01.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part B1 Second Line Treatment | Part B2 Second Line Treatment
Number analyzed (Participants) | 22 | 24
percentage of patients | 31.8 [13.9 to 54.9] | 37.5 [18.8 to 59.4]

19. Secondary Outcome: Part C: To Estimate the Objective Response Rate (ORR) in DKK1-high G/GEJ Adenocarcinoma Patients Treated With DKN-01 in Combination With Tislelizumab + Chemotherapy Regimen (CAPOX or mFOLFOX6) as a First-line Therapy.
Description: Objective Response Rate (ORR) is defined as the proportion of patients achieving best overall response of Complete Response (CR) or Partial Response (PR) as assessed by the investigator using RECIST v1.1. Experimental group: Sirexatamab + tislelizumab + CAPOX/FOLFOX, Control group: Tislelizumab + CAPOX/FOLFOX
Time Frame: approximately 30 months
Population: Experimental group: Sirexatamab + tislelizumab + CAPOX/FOLFOX, Control group: Tislelizumab + CAPOX/FOLFOX
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part C Control First Line Treatment | Part C Experimental First Line Treatment
Number analyzed (Participants) | 85 | 85
percentage of patients | 57.6 [46.4 to 68.3] | 60 [48.8 to 70.5]
Statistical Analysis 1: Comparison: Part C Control First Line Treatment vs Part C Experimental First Line Treatment; Test type: Superiority; p = 0.3799, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.4, 95% CI 2-sided [-12.2 to 16.9]

20. Secondary Outcome: Part C: To Estimate the Duration of Response (DoR) in DKK1-high G/GEJ Adenocarcinoma Patients Treated With DKN-01 in Combination With Tislelizumab + Chemotherapy Regimen (CAPOX or mFOLFOX6) as a First-line Therapy.
Description: The duration of response (DoR) is defined only for responders (patients with a BOR of CR or PR) at the time from initial response (CR or PR) until radiographically documented progressive disease or death due to any cause, whichever is earlier. For ORR patient without PD or death, DoR is censored at the most recent tumor assessment before the data cutoff or study withdrawal, whichever occurs first.
Time Frame: approximately 30 months
Population: Experimental group: Sirexatamab + tislelizumab + CAPOX/FOLFOX, Control group: Tislelizumab + CAPOX/FOLFOX
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part C Control First Line Treatment | Part C Experimental First Line Treatment
Number analyzed (Participants) | 49 | 51
months | 12.06 [7.56 to 16.99] | 6.24 [5.06 to 8.54]

21. Secondary Outcome: Part C: To Estimate the Overall Survival (OS) in DKK1-high G/GEJ Adenocarcinoma Patients Treated With DKN-01 in Combination With Tislelizumab + Chemotherapy Regimen (CAPOX or mFOLFOX6) as a First-line Therapy.
Description: Overall survival (OS) OS is defined as the time from the date of randomization to death due to any cause. For a patient who is not known to have died by the end of study follow-up, observation of OS is censored at the date the patient was last known to be alive (i.e., date of last contact). Patients lacking data beyond the day of randomization is censored at the date of randomization (i.e., OS duration of 1 day).
Time Frame: approximately 30 months
Population: Experimental group: Sirexatamab + tislelizumab + CAPOX/FOLFOX, Control group: Tislelizumab + CAPOX/FOLFOX
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part C Control First Line Treatment | Part C Experimental First Line Treatment
Number analyzed (Participants) | 85 | 85
months | 18.76 [14.00 to NA] — The upper confidence limit for the 50th percentile is defined as the first time at which the upper confidence limit for S(t) (based on a ln(-lnS(t)) transformation) is less than or equal to 1-50/100 =0.5. There is never an observed failure time for which the upper bound of the confidence interval for the KM estimate (calculated using the Greenwood's method, which is different from the ln(-lnS(t)) transformation above) is less than 0.5, due to lack of events and sample size. | 15.38 [13.40 to 19.45]

22. Secondary Outcome: Part C: Assess Whether the Addition of DKN-01 With Tislelizumab + Chemotherapy Regimen (CAPOX or mFOLFOX6) Improves PFS in Patients w/ Combined Positive Score (CPS) ≥5 or CPS <5 Advanced DKK1-high and Overall G/GEJ Adenocarcinoma as a First-line Therapy.
Description: as for outcome 2
Time Frame: approximately 30 months
Population: Intent-to-Treat (ITT): All patients randomized to treatment. Patients will be included in the treatment group assigned at randomization regardless of the actual treatment received. Experimental: DKK1+tislelizumab+(CAPOX/mFOLFOX6), Control: tislelizumab+(CAPOX/mFOLFOX6).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- PFS DKK1-high Patients, Part C Experimental: Part C experimental patients will receive DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  * DKN-01 600mg: Administered by IV infusion
  * DKN-01 400mg: Administered by IV infusion
  * Tislelizumab 200mg: Administered by IV infusion
  * Tislelizumab 400mg: Administered by IV infusion
  * Oxaliplatin: Administered by IV infusion
  * Capecitabine 1000mg/ m2 BID: Administered orally
  * Leucovorin Calcium: Administered by IV infusion
  * Fluorouracil: Administered by IV infusion
- PFS DKK1-high Patients, Part C Control; PFS All Patients, Part C Control: Part C control patients will receive only tislelizumab in combination with chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  * Tislelizumab 200mg: Administered by IV infusion
  * Tislelizumab 400mg: Administered by IV infusion
  * Oxaliplatin: Administered by IV infusion
  * Capecitabine 1000mg/ m2 BID: Administered orally
  * Leucovorin Calcium: Administered by IV infusion
  * Fluorouracil: Administered by IV infusion
- PFS All Patients, Part C Experimental: Part C experimental patients will receive DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  * DKN-01 600mg: Administered by IV infusion
  * DKN-01 400mg: Administered by IV infusion
  * Tislelizumab 200mg: Administered by IV infusion
  * Tislelizumab 400mg: Administered by IV infusion
  * Oxaliplatin: Administered by IV infusion
  * Capecitabine 1000mg/ m2 BID: Administered orally
  * Leucovorin Calcium: Administered by IV i
Arm/Group | PFS DKK1-high Patients, Part C Experimental | PFS DKK1-high Patients, Part C Control | PFS All Patients, Part C Experimental | PFS All Patients, Part C Control
Number analyzed (Participants) | 22 | 22 | 85 | 85
Months | 7.43 [5.65 to 7.75] | 11.14 [7.46 to 14.42] | 7.66 [6.87 to 9.49] | 10.41 [7.75 to 13.86]
Statistical Analysis 1: Comparison: PFS DKK1-high Patients, Part C Experimental vs PFS DKK1-high Patients, Part C Control; Test type: Superiority; p = 0.8679, Log Rank; Stratified Log-rank Test
Statistical Analysis 2: Comparison: PFS All Patients, Part C Experimental vs PFS All Patients, Part C Control; Test type: Superiority; p = 0.9676, Log Rank; Stratified Log-rank Test
Statistical Analysis 3: Comparison: PFS DKK1-high Patients, Part C Experimental vs PFS DKK1-high Patients, Part C Control; Test type: Superiority; Hazard Ratio (HR) = 1.50, 95% CI 2-sided [0.74 to 3.05]
Statistical Analysis 4: Comparison: PFS All Patients, Part C Experimental vs PFS All Patients, Part C Control; Test type: Superiority; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.98 to 2.05]

23. Secondary Outcome: Part C: To Assess Whether the Addition of DKN-01 With Tislelizumab + Chemotherapy Regimen (CAPOX or mFOLFOX6) Improves ORR in Patients With CPS ≥5 or CPS <5 Advanced DKK1-high and Overall G/GEJ Adenocarcinoma as a First-line Therapy.
Description: Objective Response Rate (ORR) is defined as the proportion of patients achieving best overall response of Complete Response (CR) or Partial Response (PR) as assessed by the investigator using RECIST v1.1. Risk difference (RD)(%) or ORR: Positive RD implies the exposure is associated with a higher probability of the outcome occurring. Negative RD indicates the exposure is associated with a lower probability of the outcome occurring.
Time Frame: approximately 30 months
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- ORR DKK1-high Patients, Part C Experimental; ORR All Patients, Part C Experimental: Part C experimental patients will receive DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  * DKN-01 600mg: Administered by IV infusion
  * DKN-01 400mg: Administered by IV infusion
  * Tislelizumab 200mg: Administered by IV infusion
  * Tislelizumab 400mg: Administered by IV infusion
  * Oxaliplatin: Administered by IV infusion
  * Capecitabine 1000mg/ m2 BID: Administered orally
  * Leucovorin Calcium: Administered by IV infusion
  * Fluorouracil: Administered by IV infusion
- ORR DKK1-high Patient, Part C Control; ORR All Patients, Part C Control: Part C control patients will receive only tislelizumab in combination with chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  * Tislelizumab 200mg: Administered by IV infusion
  * Tislelizumab 400mg: Administered by IV infusion
  * Oxaliplatin: Administered by IV infusion
  * Capecitabine 1000mg/ m2 BID: Administered orally
  * Leucovorin Calcium: Administered by IV infusion
  * Fluorouracil: Administered by IV infusion
Arm/Group | ORR DKK1-high Patients, Part C Experimental | ORR DKK1-high Patient, Part C Control | ORR All Patients, Part C Experimental | ORR All Patients, Part C Control
Number analyzed (Participants) | 16 | 14 | 51 | 49
percentage | 72.7 [49.8 to 89.3] | 63.6 [40.7 to 82.8] | 60 [48.8 to 70.5] | 57.6 [46.4 to 68.3]
Statistical Analysis 1: Comparison: ORR DKK1-high Patients, Part C Experimental vs ORR DKK1-high Patient, Part C Control; Test type: Superiority; p = 0.2649, Mantel Haenszel; Risk Difference (RD) = 8.4, 95% CI 2-sided [-18.4 to 33.6] — Common Risk Difference and 95% CI: estimated by stratified Newcombe method, weighted by minimum risk
Statistical Analysis 2: Comparison: ORR All Patients, Part C Experimental vs ORR All Patients, Part C Control; Test type: Superiority; p = 0.379, Mantel Haenszel; Risk Difference (RD) = 2.4, 95% CI 2-sided [-12.2 to 16.9]

24. Secondary Outcome: Part C: Number of Patients With Toxicity ≥Grade 3 Treatment-related Adverse Events (TRAE) Associated With Each of the Treatment Arms.
Description: To characterize the frequency of toxicity ≥Grade 3 treatment-related adverse events (TRAE) associated with each treatment arm: Control (tislelizumab in combination with chemotherapy regimen (CAPOX or mFOLFOX6) and Experimental (DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6))
Time Frame: approximately 30 months
Population: 170 patients were randomized and 169 patients were treated with study medication: 84 in the Experimental group and 85 in the Control group.
Measure: Number; unit: number of patients
Groups:
- Part C Control First Line Treatment: Part C control patients will receive only tislelizumab in combination with chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  * Tislelizumab 200mg: Administered by IV infusion
  * Tislelizumab 400mg: Administered by IV infusion
  * Oxaliplatin: Administered by IV infusion
  * Capecitabine 1000mg/ m2 BID: Administered orally
  * Leucovorin Calcium: Administered by IV infusion 8Fluorouracil: Administered by IV infusion
- Part C Experimental First Line Treatment: Part C experimental patients will receive DKN-01 in combination with tislelizumab and chemotherapy regimen (CAPOX or mFOLFOX6). Part C is restricted to patients who have not had prior systemic therapy for locally advanced or metastatic disease. Patients may have received prior neoadjuvant or adjuvant therapy as long as it was completed without disease recurrence for at least 6 months.
  * DKN-01 600mg: Administered by IV infusion
  * DKN-01 400mg: Administered by IV infusion
  * Tislelizumab 200mg: Administered by IV infusion
  * Tislelizumab 400mg: Administered by IV infusion
  * Oxaliplatin: Administered by IV infusion
  * Capecitabine 1000mg/ m2 BID: Administered orally
  Leucovorin Calcium: Administered by IV infusion
  Fluorouracil: Administered by IV infusion
Arm/Group | Part C Control First Line Treatment | Part C Experimental First Line Treatment
Number analyzed (Participants) | 85 | 84
number of patients | 53 | 57

ADVERSE EVENTS:
Time Frame: Up to 30 months
Arm/Group | Part A First Line Treatment | Part B1 Second Line Treatment | Part B2 Second Line Treatment | Part C Control First Line Treatment | Part C Experimental First Line Treatment
All-Cause Mortality (participants affected / at risk) | 18/25 | 14/24 | 16/28 | 48/85 | 38/85
Serious Adverse Events (participants affected / at risk) | 11/25 | 13/24 | 13/28 | 33/85 | 37/85
Other Adverse Events (participants affected / at risk) | 25/25 | 23/24 | 24/28 | 82/85 | 83/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A First Line Treatment (N=25) | Part B1 Second Line Treatment (N=24) | Part B2 Second Line Treatment (N=28) | Part C Control First Line Treatment (N=85) | Part C Experimental First Line Treatment (N=85)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Eosinophilic myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 1
Ophthalmoplegia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 4 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Entercolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 1 | 6 | 3
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 3
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Hemoglobin decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 5 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A First Line Treatment (N=25) | Part B1 Second Line Treatment (N=24) | Part B2 Second Line Treatment (N=28) | Part C Control First Line Treatment (N=85) | Part C Experimental First Line Treatment (N=85)
Nausea (Gastrointestinal disorders) | 19 | 7 | 5 | 27 | 31
Diarrhoea (Gastrointestinal disorders) | 18 | 4 | 0 | 23 | 23
Constipation (Gastrointestinal disorders) | 12 | 5 | 1 | 30 | 21
Vomiting (Gastrointestinal disorders) | 11 | 3 | 2 | 17 | 22
Abdominal pain (Gastrointestinal disorders) | 6 | 8 | 5 | 18 | 10
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 14 | 10
Dry mouth (Gastrointestinal disorders) | 5 | 2 | 0 | 4 | 5
Dysphagia (Gastrointestinal disorders) | 4 | 0 | 2 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 11 | 7
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 6 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 6 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral discharge (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 10 | 1 | 0 | 37 | 31
Platelet count decreased (Investigations) | 7 | 0 | 1 | 34 | 18
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 3 | 21 | 14
Weight decreased (Investigations) | 5 | 2 | 0 | 13 | 16
Blood bilirubin increased (Investigations) | 4 | 3 | 5 | 9 | 5
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 14 | 11
Lymphocyte count decreased (Investigations) | 3 | 2 | 1 | 2 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 9 | 4
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 6 | 0
Troponin T increased (Investigations) | 2 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 7
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 1 | 3 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 3 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 2 | 2
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 3 | 2
Human chorionic gonadotropin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 2 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 4 | 4 | 30 | 26
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2 | 3 | 6 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 5 | 3 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4 | 2 | 5 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 8 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0
Food aversion (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 0 | 0 | 32 | 35
Neuropathy peripheral (Nervous system disorders) | 4 | 0 | 0 | 15 | 21
Headache (Nervous system disorders) | 7 | 0 | 1 | 8 | 11
Dizziness (Nervous system disorders) | 4 | 0 | 1 | 10 | 6
Dysgeusia (Nervous system disorders) | 4 | 0 | 0 | 6 | 4
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 8 | 5
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 2 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0 | 2 | 2
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vocal cord paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 17 | 7 | 6 | 23 | 25
Oedema peripheral (General disorders) | 6 | 2 | 2 | 5 | 7
Pyrexia (General disorders) | 2 | 3 | 0 | 21 | 13
Asthenia (General disorders) | 2 | 1 | 1 | 9 | 9
Mucosal inflammation (General disorders) | 3 | 2 | 0 | 4 | 9
Chills (General disorders) | 3 | 1 | 1 | 6 | 2
Temperature intolerance (General disorders) | 4 | 0 | 0 | 2 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 1
Medical device pain (General disorders) | 1 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 3 | 3
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 1
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Medical device site erosion (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 2 | 3
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 1 | 0 | 1 | 1
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site rash (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 | 0 | 0 | 17 | 17
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 7 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 9 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2 | 0 | 4 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 4 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 11 | 4
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0 | 11 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 8 | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 5 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 6 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1 | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 6 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 6 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 3 | 0 | 3 | 7 | 6
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 7 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 6 | 1
Oral candidiasis (Infections and infestations) | 2 | 0 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 6
Otitis media (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2 | 2
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 1 | 4
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Penile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 6 | 3 | 24 | 22
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 6 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Iron deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 14 | 7
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 3 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 1 | 3 | 1
Visual impairment (Eye disorders) | 3 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 2 | 1 | 0 | 0 | 2
Dermatochalasis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 2 | 2
Retinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 1
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 2 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1
Hyalosis asteroid (Eye disorders) | 0 | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal drusen (Eye disorders) | 0 | 0 | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 3 | 3 | 2 | 4
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 1 | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 3 | 1
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 1 | 3 | 8 | 6
Depression (Psychiatric disorders) | 2 | 2 | 1 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 2 | 3
Mental status changes (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Adjustment disorder with anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 3 | 1 | 2 | 2 | 5
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 2 | 3
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 5 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 2 | 2
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to lack of efficacy. Therefore, only limited efficacy analyses were performed on the primary and limited secondary efficacy endpoints. Parts A+B were initiated and completed. Part C was initiated upon completion of Parts A+B. Due to termination of the program during Part C, combined analysis for Parts A+B and C was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 45 days prior to submission for Publication, Institution submits proposed Publication to Sponsor. Review Period for abstracts/poster presentations is 30 days. Sponsor may notify Institution in writing that patent applications will be filed and publication may be deferred up to 60 days. If Publication has Sponsor Confidential Information (CI) & Sponsor requests Institution to delete CI, Institution agrees to delete CI if it does not preclude the accurate interpretation of Study results.

DOCUMENTS (3):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT04363801/Prot_000.pdf
  • Statistical Analysis Plan: SAP Part A+B (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT04363801/SAP_001.pdf
  • Statistical Analysis Plan: SAP Part C (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT04363801/SAP_002.pdf